CLINICAL TRIAL: NCT06988605
Title: Real-world Experience Using Nemolizumab in the Treatment of Moderate-to-Severe Atopic Dermatitis in Adolescents & Adults
Acronym: RE-UNITE AD
Status: Recruiting | Type: Observational
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: SPR207806
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nemolizumab: Participants with moderate-to-severe AD who are receiving nemolizumab (Nemluvio®) in routine clinical practice will be observed for approximately 12 months.

SUMMARY:
The main aim of the study is to assess real-world effectiveness of nemolizumab in Atopic Dermatitis (AD) as measured by physician assessment and patient reported outcome (PRO) in clinical practice at Month 6.

DETAILED DESCRIPTION:
This prospective, multicenter, non-interventional study (NIS) seeks to evaluate treatment with nemolizumab of moderate-to-severe AD in adolescents and adults over an approximately 12-month period using physician assessments in routine clinical practice and PRO measures.

Treatment with nemolizumab will be determined solely by the participant's physician prior to study enrollment. No additional visits, procedures, or laboratory tests are required outside of routine clinical practice. The visit structure is not defined by the study protocol but is determined by routine medical practice. The visit schedule is intended to facilitate a systematic data assessment according to clinical routine. A sub-study will be completed in Germany and the UK at selected sites in which participants will complete the Peak Pruritus (PP) Numerical Rating Scale (NRS), Average Pruritus (AP) NRS, Sleep Disturbance (SD) NRS, and Pain NRS on a daily basis from Day -1 to Day 14. Data collection will occur remotely, and no clinic visits will be required.

ELIGIBILITY:
Inclusion Criteria:

* Participants who, according to the treating physician's decision and in line with the local package label, start treatment with nemolizumab (Nemluvio®).
* Adolescent and adult participants aged >=12 years with moderate-to-severe AD.
* Participants who signed the written informed consent form (ICF) or had it signed by their legal representative.

Exclusion Criteria:

* Have contraindication(s) for the use of nemolizumab (Nemluvio®) according to the local package label.
* Participants who received treatment with a drug under clinical development/investigation within 3 months prior to baseline.
* Participants who received nemolizumab previously.
* Participants who are mentally, physically, or linguistically unable to understand the content of the ICF and/or to complete the study questionnaires.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The clinical decision for treatment with nemolizumab has to be made by the physicians independently of the participation in this NIS and prior to the informed consent process. Participants greater than or equal to (>=) 12 years of age will be eligible for the trial.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-11-06 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Investigator Global Assessment (IGA) at Month 6 | At Month 6
  The IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) used by the investigator or trained designee to evaluate the global severity of AD and the clinical response to a treatment.
Peak Pruritus Numerical Rating Scale (PP NRS) at Month 6 | At Month 6
  The PP NRS is a single question validated PRO assessment that participants will use to report the maximum intensity of their pruritus (itch). The PP NRS consists of the following question: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Here, a lower score indicates a better outcome.

SECONDARY OUTCOMES:
Eczema Area and Severity Index (EASI) up to Month 12 | Up to Month 12
  The EASI is a validated measure commonly used in clinical trials and clinical practice to assess the severity and the extent of AD signs. The EASI score is a composite score ranging from 0 to 72. The severity of erythema, induration/papulation, excoriation, and lichenification will be assessed by the investigator or trained designee on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. In addition, the extent of AD involvement in each of the 4 body areas will be assessed as a percentage by body area of head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. A higher score indicates severe AD.
Scoring Atopic Dermatitis (SCORAD) up to Month 12 | Up to Month 12
  The SCORAD is a validated measure commonly used in clinical trials and clinical practice to assess the severity and the extent of AD signs and symptoms. The SCORAD ranges from 0 to 103 and has 3 components: extent, intensity, and patient-reported symptoms of pruritus and sleep loss. The investigator or trained designee will assess the severity of 6 signs of AD (erythema, edema/papulation, oozing/crust, excoriation, lichenification, and dryness), each on a scale ranging from 0 (absence) to 3 (severe). The investigator or trained designee will also ask the participant to evaluate their symptoms of pruritus and sleep loss (average for the last 3 days/nights), each evaluated on a visual analogue scale (VAS) from 0 to 10. A higher score indicates severe AD.
Investigator Global Assessment (IGA) up to Month 12 | Up to Month 12
  The IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) used by the investigator or trained designee to evaluate the global severity of AD and the clinical response to a treatment.
Peak Pruritus Numerical Rating Scale (PP NRS) up to Month 12 | Up to Month 12
  The PP NRS is a single question validated PRO assessment that participants will use to report the maximum intensity of their pruritus (itch). The PP NRS consists of the following question: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Here, a lower score indicates a better outcome.
Average Pruritus Numerical Rating Scale (AP NRS) up to Month 12 | Up to Month 12
  The AP NRS is a single question assessment that participants will use to report the average intensity of their pruritus (itch). The AP NRS consists of the following question: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch overall during the previous 24 hours?". Here, a lower score indicates a better outcome.
Sleep Disturbance Numerical Rating Scale (SD NRS) up to Month 12 | Up to Month 12
  The SD NRS is a single-item PRO for quantifying sleep disturbance. The SD NRS consists of the following question: "On a scale of 0 to 10, with 0 being 'no sleep loss related to the symptoms of my skin disease (atopic dermatitis)' and 10 being 'I did not sleep at all due to the symptoms of my skin disease (atopic dermatitis)', how would you rate your sleep last night?". Here, a lower score indicates a better outcome.
Pain Numerical Rating Scale (Pain NRS) up to Month 12 | Up to Month 12
  The Pain NRS is a single-item assessment with a potential follow-up question that participants will use to report the average intensity of their pain. The Pain NRS consists of the following question: "Over the past 24 hours, how severe was the pain in your skin?". If the participant rates their pain from 1 to 10, then the following question will be asked: "Do you think the pain is part of the itch, from scratching or both?". Here, a lower score indicates a better outcome.

CONTACTS AND LOCATIONS:
Locations (110):
- United States (62):
  - Galderma Investigational Site - 8893, Birmingham, Alabama
  - Galdrma Investigational Site - 7077, Phoenix, Arizona
  - Galderma Investigational Site 7060, Phoenix, Arizona
  - Galderma Investigational Site - 8535, Phoenix, Arizona
  - Galderma Investigational Site - 7067, Tucson, Arizona
  - Galderma Investigational Site - 7074, Corona, California
  - Galderma Investigational Site 6836, Fountain Valley, California
  - Galderma Investigational Site 8224, Fremont, California
  - Galderma Investigational Site 7100, Irvine, California
  - Galderma Investigational Site 7099, Los Angeles, California
  - Galderma Investigational Site 8553, Newport Beach, California
  - Galderma Investigational Site 6836, San Francisco, California
  - Galderma Investigational Site, Santa Monica, California
  - Galderma Investigational Site 7107, Thousand Oaks, California
  - Galderma Investigational Site 7061, Castle Rock, Colorado
  - Galderma Investigational Site 7059, Fairfield, Connecticut
  - Galderma Investigational Site 7105, Coral Gables, Florida
  - Galderma Investigational Site 7063, Cutler Bay, Florida
  - Galderma Investigational Site 7101, Jupiter, Florida
  - Galderma Investigational Site 7021, Miami, Florida
  - Galderma Investigational Site 7084, Miami, Florida
  - Galderma Investigational Site 7078, Miami, Florida
  - Galderma Investigational Site 7070, North Miami Beach, Florida
  - Galderma Investigational Site 7090, St. Petersburg, Florida
  - Galderma Investigational Site 7054, Tampa, Florida
  - Galderma Investigational Site 7091, Tampa, Florida
  - Galderma Investigational Site 7058, Chicago, Illinois
  - Galderma Investigational Site 8142, Indianapolis, Indiana
  - Galderma Investigational Site 7083, West Lafayette, Indiana
  - Galderma Investigational Site 7098, Columbia, Maryland
  - Galderma Investigational Site 8012, Glenn Dale, Maryland
  - Galderma Investigational Site 7068, Rockville, Maryland
  - Galderma Investigational Site 7065, Brighton, Massachusetts
  - Galderma Investigationa Site 7104, Milford, Massachusetts
  - Galderma Investigational Site 7066, Auburn Hills, Michigan
  - Galderma Investigational Site 7071, Caledonia, Michigan
  - Galderma Investigational Site 7108, Grandville, Michigan
  - Galderma Investigational Site 7072, Troy, Michigan
  - Galderma Investigational Site 7057, Lee's Summit, Missouri
  - Galderma Investigational Site 7076, St Louis, Missouri
  - Galderma Investigational Site 8848, Las Vegas, Nevada
  - Galderma Investigational Site 7055, Portsmouth, New Hampshire
  - Galderma Investigational Site - Site 7080, Auburn, New York
  - Galderma Investigational Site # 7052, East Syracuse, New York
  - Galderma Investigational Site - 8282, Mount Kisco, New York
  - Galderma Investigational Site - 7051, New York, New York
  - Galderma Investigational Site 7109, New York, New York
  - Galderma Investigational Site 8279, New York, New York
  - Galderma Investigational Site 7081, Dayton, Ohio
  - Galderma Investigational Site 7073, Gresham, Oregon
  - Galderma Investigational Site 8559, Philadelphia, Pennsylvania
  - Galderma Investigational Site 7103, Philadelphia, Pennsylvania
  - Galderma Investigational Site 7106, Bluffton, South Carolina
  - Galderma Investigational Site 7082, Cedar Park, Texas
  - Galderma Investigational Site 8238, Dallas, Texas
  - Galderma Investigational Site 7062, Edinburg, Texas
  - Galderma Investigational Site 7088, Grapevine, Texas
  - Galderma Investigational Site 7102, Houston, Texas
  - Galderma Investigational Site 7069, Sugar Land, Texas
  - Galderma Investigational Site 8618, Waco, Texas
  - Galderma Investigational Site 7085, Bountiful, Utah
  - Galderma Investigational Site 7079, Vienna, Virginia
- Germany (25):
  - Galderma Investigational Site 6374, Karlsruhe, Baden-Wurttemberg
  - Galderma Investigational Site 6412, Langenau, Baden-Wurttemberg
  - Galderma Investigational Site 6416, Augsburg, Bavaria
  - Galderma Investigational Site 6369, Erlangen, Bavaria
  - Galderma Investigational Site 6417, Regensburg, Bavaria
  - Galderma Investigational Site 6419, Remscheid, North Rhine-Westphalia
  - Galderma Investigational Site 6387, Ahaus
  - Galderma Investigational Site 6383, Augsburg
  - Galderma Investigational Site 6385, Berlin
  - Galderma Investigative Site 6172, Berlin
  - Galderma Investigational Site 6366, Berlin
  - Galderma Investigational Site 6398, Bernau bei Berlin
  - Galderma Investigational Site 6386, Bielefeld
  - Galderma Investigational Site 6066, Buxtehude
  - Galderma Investigational Site 6414, Gladbeck
  - Galderma Investigational Site 6418, Großenhain
  - Galderma Investigational Site 6370, Haslach im Kinzigtal
  - Galderma Investigational Site 6420, Hersbruck
  - Galderma Investigational Site 6384, Koblenz
  - Galderma Investigational Site 6013, Lübeck
  - Galderma Investigational Site 6373, Mainz
  - Galderma Investigational Site 6371, Oberursel
  - Galderma Investigational Site 6411, Oranienburg
  - Galderma Investigational Site 6390, Pforzheim
  - Galderma Investigational Site 6372, Quedlinburg
- United Kingdom (23):
  - Galderma Investigational Site 5408, London, Hampshire
  - Galderma Investigational Site 6401, Southampton, Hampshire
  - Galderma Investigational Site 6399, Watford, Hertfordshire
  - Galderma Investigational Site 6400, Kings Lynn, Norfolk
  - Galderma Investigational Site 5131, Harrogate, North Yorkshire
  - Galderma Investigational Site 6389, Sheffield, South Yorkshire
  - Galderma Investigational Site 6395, London, Surrey
  - Galderma Investigational Site 6392, Birmingham, West Midlands
  - Galderma Investigational Site 6404, Leeds, West Yorkshire
  - Galderma Investigational Site 6397, York, Yorkshire
  - Galderma Investigational Site 6375, Bridgend
  - Galderma Investigational Site 6388, Epsom
  - Galderma Investigational Site 6394, Harrow
  - Galderma Investigational Site 6393, Kingston upon Thames
  - Galderma Investigational Site 6415, Liverpool
  - Galderma Investigational Site 5210, London
  - Galderma Investigational Site 6368, London
  - Galderma Investigational Site 6396, Manchester
  - Galderma Investigational Site 6402, Metropolitan Borough of Wirral
  - Galderma Investigational Site 5431, Redhill
  - Galderma Investigational Site 6403, Sandbach
  - Galderma Investigational Site 5989, Swansea
  - Galderma Investigational Site 5944, Wolverhampton

IPD SHARING:
Plan to Share IPD: No